CLINICAL TRIAL: NCT05714332
Title: Impacts of an Advanced Practice Physiotherapy Model of Care for Adults With a Peripheral Musculoskeletal Disorders Referred to an Orthropaedic Outpatient Clinic: a Prospective Observational Study
Brief Title: Impacts of an Advanced Practice Physiotherapy Model of Care for Adults With a Peripheral Musculoskeletal Disorders Referred to an Orthropaedic Outpatient Clinic
Status: Completed | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Other Study IDs: v3
Record Dates: First submitted 2022-11-07; First posted 2023-02-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-08

CONDITIONS: Musculoskeletal Disorders
Keywords: Advanced practice; Physiotherapy; Musculoskeletal disorders; Orthopedic; Observation
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Advanced practice physiotherapy and orthopedic surgeon group: Patients cared by both an advanced practice physiotherapist and an orthopedic surgeon.
  Interventions: Other: Advanced practice physiotherapy and orthopedic surgeon management
- Orthopedic surgeon only group: Patients cared only by an orthopedic surgeon.
  Interventions: Other: Orthopedic surgeon management

INTERVENTIONS:
Other: Advanced practice physiotherapy and orthopedic surgeon management — Management of their musculoskeletal condition by an advanced practice physiotherapist and an orthopedic surgeon.
  Groups: Advanced practice physiotherapy and orthopedic surgeon group
Other: Orthopedic surgeon management — Management of their musculoskeletal condition by an orthopedic surgeon.
  Groups: Orthopedic surgeon only group

SUMMARY:
The goal of this prospective observational study is to evaluate advanced practice physiotherapy and orthopedic surgeon care and clinical outcomes for new patients with a peripheral musculoskeletal disorders consulting at the orthopedic outpatient clinic of the Hôpital Jean-Talon.

The main questions it aims to answer are: 1. To describe the models of care at the Hôpital Jean-Talon orthopedic outpatient clinic; 2. To assess change in pain, disability, quality of life and pain catastrophizing at 6, 12 and 26 weeks after the initial evaluation; 3. To assess interprofessional collaboration between the advanced practice physiotherapists and orthopedic surgeons; 4. To assess patient satisfaction with care; 5. To assess waiting time before an initial consultation.

Researchers will compare patients cared in the advanced practice physiotherapy and orthopedic surgeon group and the orthopedic surgeon only group.

ELIGIBILITY:
Inclusion Criteria:

* Adults with peripheral musculoskeletal disorders
* New consultation at the Hôpital Jean-Talon orthopedic outpatient clinic
* Legally able to consent
* Understand and speak French or English
* Beneficiaries of the provincial universal health insurance coverage (RAMQ)

Exclusion Criteria:

* Patients directly referred from the emergency department (not considered as patients referred to the outpatient clinic).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with a peripheral musculoskeletal disorders
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Brief pain inventory severity | 6 weeks (change from baseline)
  Pain questionnaire (0-10; higher score=worse)
Brief pain inventory severity | 12 weeks (change from baseline)
  Pain questionnaire (0-10; higher score=worse)
Brief pain inventory severity | 26 weeks (change from baseline)
  Pain questionnaire (0-10; higher score=worse)
Brief pain inventory inventory | 6 weeks (change from baseline)
  Pain interference (disability) questionnaire (0-10; higher score=worse)
Brief pain inventory inventory | 12 weeks (change from baseline)
  Pain interference (disability) questionnaire (0-10; higher score=worse)
Brief pain inventory inventory | 26 weeks (change from baseline)
  Pain interference (disability) questionnaire (0-10; higher score=worse)

SECONDARY OUTCOMES:
Shortened Disability of the Arm, Shoulder and Hand (QuickDASH) | 6 weeks (change from baseline)
  Disability questionnaire for upper extremity disorders (0-100; higher=worse)
Shortened Disability of the Arm, Shoulder and Hand (QuickDASH) | 12 weeks (change from baseline)
  Disability questionnaire for upper extremity disorders (0-100; higher=worse)
Shortened Disability of the Arm, Shoulder and Hand (QuickDASH) | 26 weeks (change from baseline)
  Disability questionnaire for upper extremity disorders (0-100; higher=worse)
Hip disability and Osteoarthritis Outcomes Score (HOOS) | 6 weeks (change from baseline)
  Disability questionnaire for hip disorders (0-100; higher=better)
Hip disability and Osteoarthritis Outcomes Score (HOOS) | 12 weeks (change from baseline)
  Disability questionnaire for hip disorders (0-100; higher=better)
Hip disability and Osteoarthritis Outcomes Score (HOOS) | 26 weeks (change from baseline)
  Disability questionnaire for hip disorders (0-100; higher=better)
Knee injury and Osteoarthritis Outcomes Score (KOOS) | 6 weeks (change from baseline)
  Disability questionnaire for knee disorders (0-100; higher=better)
Knee injury and Osteoarthritis Outcomes Score (KOOS) | 12 weeks (change from baseline)
  Disability questionnaire for knee disorders (0-100; higher=better)
Knee injury and Osteoarthritis Outcomes Score (KOOS) | 26 weeks (change from baseline)
  Disability questionnaire for knee disorders (0-100; higher=better)
Foot and Ankle Ability Measure (FAAM) | 6 weeks (change from baseline)
  Disability questionnaire for ankle/foot disorders (0-100; higher=better)
Foot and Ankle Ability Measure (FAAM) | 12 weeks (change from baseline)
  Disability questionnaire for ankle/foot disorders (0-100; higher=better)
Foot and Ankle Ability Measure (FAAM) | 26 weeks (change from baseline)
  Disability questionnaire for ankle/foot disorders (0-100; higher=better)
EQ-5D-5L | 6 weeks (change from baseline)
  Health-related quality of life questionnaire (to be converted in QALYs 0-1; higher=better)
EQ-5D-5L | 12 weeks (change from baseline)
  Health-related quality of life questionnaire (to be converted in QALYs 0-1; higher=better)
EQ-5D-5L | 26 weeks (change from baseline)
  Health-related quality of life questionnaire (to be converted in QALYs 0-1; higher=better)
EQ-5D-VAS | 6 weeks (change from baseline)
  Health-related quality of life questionnaire (0-100; higher=better)
EQ-5D-VAS | 12 weeks (change from baseline)
  Health-related quality of life questionnaire (0-100; higher=better)
EQ-5D-VAS | 26 weeks (change from baseline)
  Health-related quality of life questionnaire (0-100; higher=better)
Pain Catastrophizing Scale (PCS) | 6 weeks (change from baseline)
  Health-related quality of life questionnaire (0-50; higher=worse)
Pain Catastrophizing Scale (PCS) | 12 weeks (change from baseline)
  Health-related quality of life questionnaire (0-50; higher=worse)
Pain Catastrophizing Scale (PCS) | 26 weeks (change from baseline)
  Health-related quality of life questionnaire (0-50; higher=worse)
Patient perceptions of team effectiveness (Patient-PTE) | 0 week (post initial consultation)
  Perceptions of team effectiveness questionnaire (24-144; higher=better)
modified validated version of the 9-item visit-specific satisfaction questionnaire (VSQ-9) | 0 week (post initial consultation)
  Patient satisfaction questionnaire (0-100; higher=better)
Modified MedRisk | 12 weeks
  Patient satisfaction questionnaire (0-100; higher=better)
Modified MedRisk | 26 weeks
  Patient satisfaction questionnaire (0-100; higher=better)
Provider perceptions of team effectiveness (Prodiver-PTE) | Through study completion (once)
  Perceptions of team effectiveness questionnaire (26-156; higher=better)
Waiting time | Pre-intervention
  Waiting time (time in days and minutes)
Adverse events | 12 weeks
  Rate of adverse events
Adverse events | 26 weeks
  Rate of adverse events
Treatment and compliance | 6 weeks
  Treatment received and % of treatment compliance
Treatment and compliance | 12 weeks
  Treatment received and % of treatment compliance
Treatment and compliance | 26 weeks
  Treatment received and % of treatment compliance

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche de l'Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be available upon resonable request